CLINICAL TRIAL: NCT01931995
Title: Investigation of Cortico-limbic Networks and Their Dynamics in Major Depressive Disorder
Brief Title: Investigation of Brain Network Dynamics in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Mark C. Eldaief, MD, Mark Eldaief, MD, Associate Neurologist, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2012p001784
Record Dates: First submitted 2013-08-19; First posted 2013-08-30 (Estimated); Results first posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Major Depressive Disorder, Recurrent
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TMS to positively correlated DLPFC (Active Comparator): High frequency TMS to a target region of dorsolateral prefrontal cortex which is positively correlated with the subgenual cingulate cortex
  Interventions: Device: TMS positively correlated DLPFC
- TMS to negatively correlated DLPFC (Active Comparator): High frequency TMS to a target region of dorsolateral prefrontal cortex which is positively correlated with the subgenual cingulate cortex
  Interventions: Procedure: TMS to negatively correlated DLPFC

INTERVENTIONS:
Device: TMS positively correlated DLPFC — TMS, or transcranial magnetic stimulation, is a technique that is employed to non-invasively activate or suppress targeted regions of the cerebral cortex. One TMS system has been FDA approved to treat certain medically refractory forms of depression.
  Other Names: This study will employ a TMS system that includes a stimulator, TMS coil and neuronavigation system
  Arms: TMS to positively correlated DLPFC
Procedure: TMS to negatively correlated DLPFC — TMS, or transcranial magnetic stimulation, is a way of non-invasively activating or suppressing targeted regions of the cerebral cortex. One TMS system has been FDA approved to treat certain medically refractory forms of depression.
  Other Names: This study will employ a TMS system that includes a stimulator, TMS coil and neuronavigation system
  Arms: TMS to negatively correlated DLPFC

SUMMARY:
This research study is being done to gain a better understanding about brain networks that may be involved in depression. The investigators plan to examine how these networks change after the brain is stimulated with "Transcranial Magnetic Stimulation" (TMS). TMS is a way of stimulating the brain in order to mildly activate or mildly suppress different brain areas, and is used to treat some forms of depression. It is hoped that this study will facilitate learning more about the structure and function of different brain areas and the ways that they are interconnected to form networks, both in depressed people and in people without depression. In this research study, the effects of TMS will be measured by obtaining "pictures" of the brain with "Magnetic Resonance Imaging" (MRI) and with "Positron Emission Tomography" (PET). More specifically, this will be accomplished with a combined MRI and PET scanner, which is capable of simultaneously obtaining both MRI and PET images of the brain. This scanning paradigm will allow the assessment of local metabolic changes resulting from TMS (with PET images) and brain network changes resulting from TMS (with fMRI). Changes resulting from TMS between 20 subjects with depression and 20 healthy volunteers will be calculated and will form the main outcome measure.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS), when delivered to the dorsolateral prefrontal cortex (DLPFC) is a clinically effective treatment for major depressive disorder (MDD). Network models of MDD are increasingly gaining acceptance, and functional connectivity MRI (fcMRI) has revealed topographically specific aberrations in functional network architecture in MDD. And yet, despite hints that the therapeutic effects of rTMS are actuated through distributed impacts upon cortical and subcortical limbic centers, the network effects of rTMS remain mysterious. This study seeks to investigate the way rTMS to DLPFC modulates network functional connectivity between the site of stimulation and a critical limbic region, the subgenual cingulate (sgACC), and between the sgACC and other limbic regions. In this study, high frequency rTMS will be used to stimulate the left DLPFC (recapitulating the therapeutic methodology), specifically, regions of the DLPFC that are functionally correlated and anti-correlated with the sgACC. This will be accomplished in a group of patients with MDD, and in a group of carefully matched controls. These subjects will be scanned before and after rTMS is delivered, as a way of gauging its effects. The feasibility of this design was recently demonstrated by our group (Eldaief et al. PNAS 2011). Changes induced by the stimulation will be charted with a novel combined MRI-PET (Positron Emission Tomography) scanner at the MGH Martinos Center, which is capable of simultaneously recording fcMRI BOLD (Blood oxygenation level-dependent) and 18Flurodeoxyglucose (FDG) PET data. This will permit cortico-limbic networks to be characterized dynamically through (1) examination of the differential effects of stimulating two networks in the DLPFC, and (2) by tracking the dynamic interplay between rTMS induced changes in local glucose metabolism at DLPFC and sgACC on the one hand, and changes in distributed connectivity between these regions on the other. In an exploratory aim, MDD patients will return three months later (after they have undergone a non-specific treatment intervention with their psychiatric provider) for the identical rTMS/fcMRI/FDG-PET procedures. This aim will establish, as proof of principle, that treatment of MDD is associated with changes in cortico-limbic functional network architecture, and in cortico-limbic dynamics. Eventually, it is hoped that this work will lead to the emergence of aberrant cortical dynamics as a biomarker for MDD. In addition, this work might pollinate future studies which use aberrant cortical dynamics as a novel therapeutic target upon which neuromodulatory interventions might intervene.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-50
* Patients with Major Depressive Disorder, as confirmed by a referring provider, DSM-IVR criteria, and/or a Structured Clinical Interview (SCID)
* Score of ≥18 on the 24 item version of the Hamilton Depression Rating Scale (HDRS)
* Meeting criteria to safely receive fMRI scanning, PET scanning and rTMS.

Exclusion Criteria:

* Any subject who is pregnant or lactating
* Patients with bipolar disorder, schizoaffective disorder, suicidal ideation, or any history of psychosis. Concurrent anxiety disorders will be allowed.
* Any serious concurrent medical or neurological illness
* Any contraindication to receiving TMS, fMRI or PET scans including, but not limited to having: a pacemaker, metallic implants, implanted pumps, surgical aneurysm clips, history of severe head trauma, history of seizures or a first degree relative with epilepsy, been involved in a nuclear medicine study in the past 12 months, diabetes

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2013-02; Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Eldaief, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Martinos Center for Biomedical Imaging/Massachusetts General Hospital, Charlestown, Massachusetts, United States

REFERENCES:
- [Derived] Sun W, Billot A, McMains S, Rodrigues K, Braga RM, Izquierdo-Garcia D, Eldaief MC. Relationships between local metabolic activity and distributed functional connectivity in major depressive disorder. Transl Psychiatry. 2025 Dec 1. doi: 10.1038/s41398-025-03766-w. Online ahead of print. PMID 41326377

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 45 subjects were recruited between February 2013 and June 2016. All subjects were recruited in Boston, Massachusetts.
Pre-assignment Details: 45 subjects were enrolled and 37 subjects completed all three sessions. No randomization was done.
Groups:
- TMS to Positively Correlated DLPFC: Subjects first received High frequency TMS to a target region of dorsolateral prefrontal cortex which is positively correlated with the subgenual cingulate cortex
  TMS positively correlated DLPFC: TMS, or transcranial magnetic stimulation, is a technique that is employed to non-invasively activate or suppress targeted regions of the cerebral cortex. One TMS system has been FDA approved to treat certain medically refractory forms of depression.
  Following this, there was a washout period of at least 6 days, after which they received TMS to negatively correlated DLPFC.
- TMS to Negatively Correlated DLPFC: Subjects first received high frequency TMS to a target region of dorsolateral prefrontal cortex which is negatively correlated with the subgenual cingulate cortex
  TMS to negatively correlated DLPFC: TMS, or transcranial magnetic stimulation, is a way of non-invasively activating or suppressing targeted regions of the cerebral cortex. One TMS system has been FDA approved to treat certain medically refractory forms of depression.
  After a washout period of at least 6 days they received stimulation with the other treatment (TMS to positively correlated DLPFC).
Period: First Intervention (1 Day)
Arm/Group | TMS to Positively Correlated DLPFC | TMS to Negatively Correlated DLPFC
Started | 23 | 22
Completed | 19 | 18
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: Washout (at Least 6 Days)
Arm/Group | TMS to Positively Correlated DLPFC | TMS to Negatively Correlated DLPFC
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | TMS to Positively Correlated DLPFC | TMS to Negatively Correlated DLPFC
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMS to Positively Correlated DLPFC | TMS to Negatively Correlated DLPFC | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.8 (4) | 22.7 (4) | 23.9 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 17 | 16 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 37 | 37

OUTCOME MEASURES:

1. Primary Outcome: Relative Changes in Corticolimbic Functional Connectivity as a Result of TMS
Description: The primary outcome measure is the relative change in functional connectivity in prefrontal corticolimbic brain networks resulting from TMS stimulation of two nodes in the dorsolateral prefrontal cortex: one which is positively correlated to the subgenual cingulate and one which is negatively correlated to this area. Functional connectivity is a measure of correlation strength which biologically reflects correlations between low-frequency oscillations in the fMRI blood oxygenation level dependent signal. As a correlation, this ranges from -1 to 1. This is then Fisher transformed from an r value to a z value (range -2 to -2).
Time Frame: Assessed immediately following each intervention
Measure: Mean (Standard Deviation); unit: Fisher transformed z values
Arm/Group | TMS to Positively Correlated DLPFC | TMS to Negatively Correlated DLPFC
Number analyzed (Participants) | 37 | 37
Fisher transformed z values | -0.11 (0.14) | -0.19 (0.15)

2. Secondary Outcome: Changes in Local Glucose Metabolism at Corticolimbic Network Nodes
Description: This outcome measure will employ FDG PET scanning to assess changes in local glucose metabolism resulting from TMS to two dorsolateral prefrontal stimulation targets. More specially, changes in glucose metabolism will be assessed at the stimulation targets, in the subgenual cingulate and in the amygdala. This is measured in whole brain normalized standardized uptake values (wbnSUV).
Time Frame: Assessed immediately following each intervention.
Measure: Mean (Standard Error); unit: whole brain normalized suv values
Arm/Group | TMS to Positively Correlated DLPFC | TMS to Negatively Correlated DLPFC
Number analyzed (Participants) | 37 | 37
whole brain normalized suv values | -0.06 (0.02) | 0.054 (0.02)

ADVERSE EVENTS:
Time Frame: 3 years 4 months
Arm/Group | TMS to Positively Correlated DLPFC | TMS to Negatively Correlated DLPFC
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT01931995/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT01931995/SAP_001.pdf